CLINICAL TRIAL: NCT00633711
Title: Differential Effects of Chronic Treatment of OSAS by CPAP and SOMNOsmart2 on Norepinephrine and Blood Pressure
Brief Title: Effects of Obstructive Sleep Apnea Treatment by Fixed CPAP and by Auto-CPAP (Somnosmart2)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fondazione C.N.R./Regione Toscana "G. Monasterio", Pisa, Italy (Other Government)
Collaborators: Weinmann Geräte für Medizin GmbH + Co. KG (Industry)
Responsible Party: Dr Oreste Marrone, National Research Council, Inst. of Biomedicine and Molecular Immunology, Italy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CNR-IBIM-001
Record Dates: First submitted 2008-03-04; First posted 2008-03-12 (Estimated); Last update posted 2011-06-16 (Estimated); Status verified 2010-04

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: OSAS; blood pressure; sympathetic nervous system; treatment; CPAP
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- fixed CPAP (Active Comparator)
  Interventions: Device: fixed continuous positive airway pressure (CPAP)
- Auto-CPAP (Experimental): Auto-CPAP Weinmann "Somnosmart2"
  Interventions: Device: Automatic (variable, automatically controlled) pressure CPAP

INTERVENTIONS:
Device: Automatic (variable, automatically controlled) pressure CPAP — CPAP at a variable level according to instantaneous patients' needs for treatment of sleep respiratory disorders, as evaluated by machine's software.
  Home nocturnal usage. Two-month treatment.
  Other Names: Automatic CPAP "SOMNOsmart2", Weinmann, Hamburg Germany
  Arms: Auto-CPAP
Device: fixed continuous positive airway pressure (CPAP) — CPAP at a constant level, whose efficacy on respiratory disorders has been determined by nocturnal titration.
  Home nocturnal usage. Two-month treatment.
  Other Names: fixed CPAP, constant level CPAP
  Arms: fixed CPAP

SUMMARY:
The main purpose of this study is to investigate if treatment of obstructive sleep apnea syndrome (OSAS) by continuous positive airway pressure (CPAP) given by a traditional CPAP device administering a fixed air pressure, or by one automatic CPAP device ("Somnosmart2", Weinmann, Hamburg) administering variable pressures, have different effects on sympathetic nervous system tone (as reflected by urinary excretion of norepinephrine and its catabolite normetanephrine) and on blood pressure.

DETAILED DESCRIPTION:
A nocturnal home cardiorespiratory recording will performed for diagnosis of OSA. During the same night, patients will be asked to collect their urines. Twentyfour-hour ambulatory BP monitoring (ABPM) will be performed starting from the next morning. After analysis of the polygraphic recording, subjects with AHI <15 will be excluded from the study, while CPAP will be proposed as a treatment to the other patients.

Before starting treatment, a full night standard polysomnography will be performed: in subjects assigned to fixed CPAP for attended CPAP titration; in the other subjects during application of the Somnosmart2 device, to verify if obstructive events are adequately eliminated by it.

After analysis of polysomnography, patients will be given a fixed CPAP or the auto-CPAP device for nocturnal home use. Two months later, compliance to treatment will be verified measured by the in-built time counter of the devices. Then, cardiorespiratory monitoring during application of the device used for treatment, nocturnal urine collection and 24-hour ABPM will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* Obstructive sleep apnea syndrome deserving CPAP treatment

Exclusion Criteria:

* current pharmacological treatment

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2007-03; Primary Completion 2009-12 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Blood pressure and urinary catecholamines after conventional or auto-CPAP | 2 months

SECONDARY OUTCOMES:
Relationship between catecholamines / blood pressure changes and compliance to treatment | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Oreste Marrone, MD, Principal Investigator — Fondazione C.N.R./Regione Toscana "G. Monasterio", Pisa, Italy
Locations (1):
- National Research Council - Institute of Biomedicine and Molecular Immunology (CNR - IBIM), Palermo, Italy

REFERENCES:
- [Background] Patruno V, Aiolfi S, Costantino G, Murgia R, Selmi C, Malliani A, Montano N. Fixed and autoadjusting continuous positive airway pressure treatments are not similar in reducing cardiovascular risk factors in patients with obstructive sleep apnea. Chest. 2007 May;131(5):1393-9. doi: 10.1378/chest.06-2192. PMID 17494789
- [Background] Bazzano LA, Khan Z, Reynolds K, He J. Effect of nocturnal nasal continuous positive airway pressure on blood pressure in obstructive sleep apnea. Hypertension. 2007 Aug;50(2):417-23. doi: 10.1161/HYPERTENSIONAHA.106.085175. Epub 2007 Jun 4. PMID 17548722
- [Background] Alajmi M, Mulgrew AT, Fox J, Davidson W, Schulzer M, Mak E, Ryan CF, Fleetham J, Choi P, Ayas NT. Impact of continuous positive airway pressure therapy on blood pressure in patients with obstructive sleep apnea hypopnea: a meta-analysis of randomized controlled trials. Lung. 2007 Mar-Apr;185(2):67-72. doi: 10.1007/s00408-006-0117-x. Epub 2007 Mar 28. PMID 17393240
- [Background] Haentjens P, Van Meerhaeghe A, Moscariello A, De Weerdt S, Poppe K, Dupont A, Velkeniers B. The impact of continuous positive airway pressure on blood pressure in patients with obstructive sleep apnea syndrome: evidence from a meta-analysis of placebo-controlled randomized trials. Arch Intern Med. 2007 Apr 23;167(8):757-64. doi: 10.1001/archinte.167.8.757. PMID 17452537
- [Background] Parati G, Lombardi C, Narkiewicz K. Sleep apnea: epidemiology, pathophysiology, and relation to cardiovascular risk. Am J Physiol Regul Integr Comp Physiol. 2007 Oct;293(4):R1671-83. doi: 10.1152/ajpregu.00400.2007. Epub 2007 Jul 25. PMID 17652356
- [Background] Narkiewicz K, Somers VK. Sympathetic nerve activity in obstructive sleep apnoea. Acta Physiol Scand. 2003 Mar;177(3):385-90. doi: 10.1046/j.1365-201X.2003.01091.x. PMID 12609010